CLINICAL TRIAL: NCT02455791
Title: Pilot Study for Identification of Breast Cancer Patients for Potential Avoidance of Surgery: Accuracy of Image Guided Percutaneous Sampling Compared With Surgery to Evaluate Eradication of Breast Cancer After Preoperative Chemotherapy
Brief Title: Feasibility and Identification of Breast Cancer Patients for Potential Avoidance of Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-1039; NCI-2015-01221 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Triple negative breast cancer; HER2 amplified breast cancer; Ultrasound-guided biopsy; Fine needle aspirate; FNA; Core biopsy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound-Guided Biopsy of Tumor Site (Experimental): Ultrasound-guided biopsy of the tumor site performed before scheduled surgery.
  Interventions: Procedure: Ultrasound-Guided Biopsy

INTERVENTIONS:
Procedure: Ultrasound-Guided Biopsy — Ultrasound-guided biopsy of tumor site. A needle is inserted into the affected area using an ultrasound to collect cells or tissue from a tumor mass. Two (2) types of samples collected.

SUMMARY:
The goal of this clinical research study is to compare the use of an ultrasound-guided biopsy with what is found during surgery in finding evidence of the disease.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will have an ultrasound-guided biopsy of the tumor site. To perform this biopsy, a needle is inserted into the affected area using an ultrasound to collect cells or tissue from a tumor mass. The doctor will use the ultrasound to guide the needle into the area. Two (2) types of samples will be collected: a fine needle aspirate (FNA) that collects cells and a core biopsy that collects a small piece of tissue. If the tumor is not seen well by the ultrasound, the study doctor may use a mammogram to perform the biopsy.

You will then have the same planned surgery and post-operative care that you would normally have. You will sign a separate consent for your surgery.

Your medical records may be reviewed and information recorded from your routine follow-up visits in order to follow your general health and the outcome of your surgery.

Length of Study Participation:

Your active participation in this study will be finished when you have had your surgery and completed your post-operative care.

This is an investigational study. It is investigational to compare the use of an ultrasound-guided biopsy with what is found during surgery in finding evidence of the disease.

Up to 40 participants will take part on this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. >/= 18 years old
2. Histologic diagnosis of triple negative or HER2 amplified breast cancer, clinical stage T1-4, N0-3, M0/1 receiving preoperative systemic therapy and planned surgery

Exclusion Criteria:

1) N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Ultrasound-Guided FNA and Core Biopsy of Initial Breast Cancer Region Compared to Standard Surgery with Pathologic Evaluation | 1 day
  Accuracy of FNA and core biopsy determined by comparing these biopsy results to the pathologic evaluation removed during standard surgery. Estimates and 95% confidence intervals for accuracy, sensitivity, false negative rate (FNR), specificity as well as the negative predictive value (NPV) reported for FNA and core biopsy based on the exact Clopper-Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Kuerer, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Pfob A, Sidey-Gibbons C, Lee HB, Tasoulis MK, Koelbel V, Golatta M, Rauch GM, Smith BD, Valero V, Han W, MacNeill F, Weber WP, Rauch G, Kuerer HM, Heil J. Identification of breast cancer patients with pathologic complete response in the breast after neoadjuvant systemic treatment by an intelligent vacuum-assisted biopsy. Eur J Cancer. 2021 Jan;143:134-146. doi: 10.1016/j.ejca.2020.11.006. Epub 2020 Dec 8. PMID 33307491
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org